CLINICAL TRIAL: NCT03555201
Title: Efficacy of a Physiotherapy Protocol Based on Manual Therapy in Patients With Temporomandibular Disorders.
Brief Title: Efficacy of Physiotherapy in Patients With Temporomandibular Disorders.
Acronym: MT-ATM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0022
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Temporomandibular Dysfunction (TMD)
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): Protocol of soft tissue techniques
  Interventions: Other: Regular treatment control.
- Regular treatment control. (Active Comparator): Regular treatment control.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — protocol of soft tissues techniques
  Arms: Regular treatment control.
Other: Regular treatment control. — Regular treatment control.
  Arms: Manual therapy

SUMMARY:
Objective: To evaluate the efficacy of a manual therapy protocol composed of articulatory and myofascial techniques in patients with temporomandibular dysfunction (TMD).

Methods: Randomized and controlled clinical study of patients presenting TMD. The subjects will be divided into 2 groups: 1) manual therapy group; 2) control group. There will be 4 treatment sessions during 4 weeks, with evaluations before and after the study, which include: severity of dysfunction (Helkimo Index), quality of life (Short Form 36 Health Survey), pressure pain threshold (algometer) ), cervical mobility (goniometer), mouth opening (caliper), pain intensity (Visual Analogue Scale) and cervical disability (Neck Disability Index).

DETAILED DESCRIPTION:
Introduction. Temporomandibular dysfunction (TMD) is the set of clinical manifestations that affect this joint, the masticatory muscles and the structures associated with and involved in TMJ movements. This dysfunction represents a subclassification of musculoskeletal disorders, and presents with different symptoms and signs that include pain in the jaw joint or in the tissues that surround it, generalized myofascial pain, crackling or crackling joint noise associated with the movement, decrease in joint range, functional limitation, and deviation to the opening of the jaw.

Objective. The main objective of this study is to compare the efficacy of a myofascial soft tissue treatment versus a control group in people diagnosed with TMD of myofascial origin.

Material and methods

Sample. Subjects with dagnosis of TMD according to the diagnostic criteria for the investigation of temporomandibular disorders.

Study design. Randomized clinical trial with 2 groups: Group 1. Manual therapy protocol of SOFT TISSUES; Group 2. Regular treatment control.

Evaluations. Clinical interview with anthropometric data and characteristics of the pathology.

There will be 3 evaluations: at the beginning of the study, at the end of the treatment (at 4 weeks) and at 8 weeks as part of the follow-up period.

In addition, it includes the following evaluation instruments:

* Visual Analog Scale (EVA)
* Algometry of the masseter, temporal and ECOM muscles.
* Oral opening range.
* Range of cervical joint movement.
* Quality of life questionnaire related to oral health OHIP-14.
* Quality of life questionnaire SF-36.
* Index of clinical dysfunction of Helkimo.
* Cervical disability index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMD or myofascial pain according to the Helkimo index.
* Use of the discharge splint, except in the 2 weeks prior to the study.
* Age of the subjects between 18 and 65 years old.
* Presence of TMD signs and symptoms in the 3 months prior to the study, such as limitations in movements, pain and / or deviation during opening of the mouth, muscular sensitivity, and sounds produced by the joint during opening of the mouth.
* Limitation of active vertical opening of the mouth <40 mm.
* Bilateral pain that surrounds the areas of the temporal and the masseter.
* Presence of at least one trigger point in the masseter and temporal muscles.
* Patients who sign the informed consent.

Exclusion Criteria:

* That they did not use the splint, except in the 2 weeks prior to the study.
* Presence of systemic, rheumatic or central nervous system diseases.
* Trauma or previous surgical intervention in the ATM region.
* History of some type of treatment (physiotherapy or acupuncture) in the 3 months prior to the study.
* Use of analgesics or muscle relaxants at least 24 hours before the evaluations and during the treatment period.
* Presence of another type of orofacial pain disorder.
* Presence of signs or symptoms of disc displacement, osteoarthritis or TMJ arthritis.
* Positive extension-rotation test (vertebral artery test or Klein test) or cerebrovascular changes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | 8 weeks
  Pain intensity scale. This scale consists of a horizontal line of 100 mm, delimited at one end by 0 mm (no pain) and at the other end by 100 mm (worst pain imaginable). This scale has shown a high validity and reliability for the assessment of the pain intensity of the patient

SECONDARY OUTCOMES:
Severity and degree of dysfunction | 8 weeks
  Helkimo Index. This index is based on the evaluation of five clinical signs: 1. Alteration of the range of movement by measuring the amplitude of the movements of the jaw: opening, lateralisation and protrusion of the jaw; 2. Alteration of the TMJ function (appearance of sounds in the joint during the vertical opening of the mouth, and mandibular trajectory pattern); 3. Muscle pain; 4. Pain upon palpation of the TMJ; 5. Pain during the movement of the jaw38. Each item evaluated is scored with values of 0, 1 or 5, with the sum of the scores of the clinical signs evaluated, the one referring to describing the severity and the group for each patient with TMD41. If the score obtained is 0, patients are included in group 0 (absence of symptoms). Scores from 1 to 4, group 1 (mild dysfunction). Scores from 5 to 9, group 2 (moderate dysfunction). And finally, if the score is from 10 to 25, the patients belong to group 3 (severe dysfunction).
Health status | 8 weeks
  Quality of life questionnaire. The SF-36v2 is composed of 36 items with Likert type response options, which are included in 8 dimensions: Physical Function (FF, 10 items), Physical Role (RF, 4 items), Body Pain (DC, 2 items) , General Health (SG, 6 items), Vitality (VT, 4 items), Social Function (FS, 2 items), Emotional Role (SR, 3 items) and Mental Health (SM, 5 items). The scores range from 0 to 100 in each dimension, with the highest scores associated with a better state of health. This questionnaire has demonstrated a high internal consistency with a Cronbach's alpha value of more than 0.70, and an adequate reliability (ICC = 0.73-0'86).
Cervical disability | 8 weeks
  Cervical disability questionnaire (NDI). It is a self-completed questionnaire formed by 10 sections: cervical pain intensity, personal care, weight lifting, reading, headache, concentration ability, work capacity, driving, sleep and leisure activities. The scores for each section range from 0 to 5, being 0 (without disability) and 5 (total disability). If a score ranges from 0 to 4, the patient would not have cervical disability. Scores from 5 to 14 (mild disability), from 15 to 24 (moderate disability), from 25 to 34 (severe disability) and from 35 to 50 (complete disability). Therefore, the maximum score that can be reached in this questionnaire is 509.45. The test-retest reliability has been shown to be optimal with an intraclass correlation coefficient of 0.978, and a high internal consistency with a Cronbach's alpha coefficient of 0.937.
Opening range of the mouth | 8 weeks
  Vernier caliper. To measure the active opening of the mouth without pain a vernier caliper will be used (Vernier Caliper). To do this, patients remain in a sitting position and are asked to perform a maximum opening of the mouth without pain. The distance between the upper and lower central incisors of the mandible is measured, using the millimeters as the unit of measurement. 3 consecutive measurements are made with rest intervals of 30 seconds. The final measurement is obtained based on the average of the 3 results belonging to the previous measurements. This procedure has shown high intra-rater reliability (ICC = 0'9-0'98).
Pressure pain threshold | 8 weeks
  Algometer. To assess the pain threshold at the pressure of the masseter, temporal and ECOM muscles, a mechanical pressure algometer (Wagner Instruments FDK 20) will be used. The pressure pain threshold is the minimum pressure that is needed to cause pain or discomfort at a certain point. In obtaining the result, the average of the 3 scores obtained from each point was made. The reliability of this procedure is high in healthy subjects [BCI = 0.91 (95% confidence interval: 0.82-0.97)] 28.31. In patients with TMD, reliability is moderate (ICC = 0.64)
Cervical mobility | 8 weeks
  Goniometer. The range of joint movement of the neck is measured by the use of a goniometer. Flexion, extension, lateral tilt and cervical rotation are assessed. To be able to perform the measurement, the patient is asked to remain in a sitting position keeping his back at 90 degrees and his head in a neutral position. The physiotherapist instructs the patients to perform the previously explained movements, until reaching the maximum range of movement or in the presence of pain. We proceed to evaluate mobility in the 3 planes: sagittal plane, frontal plane and transverse plane. 3 measurements of each movement are made, and the final measurement obtained is the average of each previous result.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Valencia, Spain